CLINICAL TRIAL: NCT06231108
Title: "Assessment of the Short Effects of Taping on the Foot, Knee, and Hip Regions on Balance Skills in Children With Mildly Affected Cerebral Palsy"
Brief Title: Which Taping Technique is More Effective on Balance Skills in Children With Mildly Affected Cerebral Palsy?
Status: Recruiting | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Seda AYAZ TAŞ, Assistant Professor, Abant Izzet Baysal University
Other Study IDs: BAIBU-FTR-SAT-3
Record Dates: First submitted 2024-01-21; First posted 2024-01-30 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Balance, Postural; Kinesio Tape
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case Group: "In the Single Group, three different taping applications will be performed."
  Interventions: Other: Kinesio Taping

INTERVENTIONS:
Other: Kinesio Taping — "Three different taping applications will be applied, namely ankle correction, quadriceps facilitation, and gluteus maximus facilitation."
  1. Taping: Functional correction technique will be used to facilitate dorsal flexion movement."
  2. Taping: Quadriceps Femoris (QF) Facilitation Technique - In taping to activate the QF muscle and regulate muscle tone, the patient will be placed in a supine position with hips and knees in neutral.
  3. Taping: Gluteus Maximus (GM) Facilitation Technique - For taping to facilitate the GM muscle, a double-band application will be performed.

SUMMARY:
"Our study aims to determine which of ankle correction, quadriceps facilitation, and gluteus maximus facilitation taping provides a better immediate effect on balance skills in children with mildly affected cerebral palsy. Children whose parents have given consent for the study will undergo three different taping applications with a one-week interval. After each taping application, a 15-minute waiting period will be observed, followed by balance assessment using the Wii Balance System with eyes open and closed."

DETAILED DESCRIPTION:
"Our study aims to investigate which of ankle taping, quadriceps femoris facilitation taping, and gluteus maximus facilitation taping is more effective on balance skills in children with mildly affected cerebral palsy. The study will invite ambulatory children aged 4-15 receiving special education and rehabilitation support at the Turkish Spastic Children Foundation, and those who agree to participate will be included. First, the demographic data of the children will be recorded, and then they will be assessed using the Gross Motor Function Classification System, Eating and Drinking Abilities Classification System, Hand Skills Classification System, and Communication Function Classification System.

Each child will undergo three different taping applications with a one-week interval. After each taping application, a 15-minute wait period will be observed, followed by static balance measurement using the Wii Balance Board with eyes open and closed, and the results will be recorded. SPSS (Statistical Package for Social Sciences) version 20.0 will be used for the statistical analysis of the data. The Shapiro-Wilk test will be used to determine the normality of data distributions. Parametric tests will be employed for data showing normal distribution, while non-parametric tests and one-way analysis of variance (ANOVA) will be used for data not showing normal distribution. If subgroup analysis of demographic data and clinical characteristics of cases is needed, the Independent Sample T-test or Mann-Whitney U test, and Chi-square test will be used.

To determine the relationship between independent variables, either Pearson correlation test or Spearman correlation test will be selected based on the normality of data distribution. A significance level of p < 0.05 will be considered statistically significant in all analyses. The results of the research aim to reveal which taping technique is more effective on balance skills and to promote the widespread use of the more effective technique in clinical practice."

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of bilateral spastic type cerebral palsy (CP),
* Age between 4-15 years,
* Communication Function Classification System (CFCS) level 1-2,
* Gross Motor Function Classification System (GMFCS) level 1-2,
* Volunteering to participate in the study.

Exclusion criteria:

* Having experienced lower extremity fracture, muscle-tendon, or bone surgery in the last 6 months, or undergone spine or orthopedic surgery that would affect the lower extremity,
* Exposure to any pharmacological agent or intervention inhibiting spasticity in the last 6 months,
* Developing an allergic reaction to kinesio tape."

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: "Cooperative children diagnosed with mild cerebral palsy with GMFCS levels 1 and 2."
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2024-01-21 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Static Balance Assessment | day 1
  Wii Balance Board, which has become an alternative for balance measurement due to its portability and low cost compared to specialized laboratory environments and complex devices. The Wii Balance Board transmits the vertical ground reaction forces generated at the four corners when an individual is on the device to the Wii system via Bluetooth.To assess static balance in the participating children, the Fizyosoft Balance System developed by engineers and physiotherapists will be used.Children will be instructed to place their feet parallel to each other on the device and remain motionless for up to 15 seconds with eyes open and closed during the measurement. The coordinate values of the individuals' body weight center will be recorded in centimeters, while the performance value will be stored in the system as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Ozge KARANLIK, Msc, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu Abant Izzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No